CLINICAL TRIAL: NCT06659354
Title: Targeting Health and Resilience for Individuals With a Vulnerable Eating History (THRIVE)
Brief Title: Preventing Disordered Eating and Body Dissatisfaction Among High-risk Pregnant Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Vanderkruik, Associate Director of Research and Cognitive Behavioral Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023P000630
Record Dates: First submitted 2024-10-18; First posted 2024-10-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Eating Disorders; Body Dissatisfaction
Keywords: Eating Disorder; Body Dissatisfaction; Body Image; Pregnancy
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant Body Project (PBP) (Experimental): The Body Project is typically delivered as four 1-hour weekly sessions consisting of written, verbal, and behavioral exercises. The sessions aim to induce cognitive dissonance by encouraging participants to challenge the thin-ideal, a theoretically and empirically supported component of ED prevention. This adapted version of the Body Project (the Pregnant Body Project; PBP) consists of 6 1-hour, weekly group sessions delivered via Zoom. Since the target population consists of individuals with histories of an ED or disordered eating behaviors, PBP also includes elements from a treatment intervention (i.e., the Body Project Treatment 8.0 manual). PBP was adapted iteratively with a needs assessment, expert stakeholder input, and participant feedback following a mock trial with individuals with lived experience (i.e., individuals with histories of an ED who have given birth). This condition will be peer-delivered by facilitators with lived experience.
  Interventions: Behavioral: Pregnant Body Project (PBP)
- Pregnancy Health Education (PHE) (Placebo Comparator): This time- dose- and attention- matched control condition accounts for the potential effects of time spent and support from group members and facilitators. Participants assigned to the PHE group will also be asked to attend 6, 1-hour, weekly group sessions via Zoom. During the sessions participants receive psychoeducation on body image and disordered eating during pregnancy but will not engage in any dissonance-inducing exercises. Participants will also receive lifestyle education specific to pregnancy (e.g., proper nutrition, sleep, physical activity), tied back to body image and disordered eating.
  Interventions: Behavioral: Pregnancy Health Education (PHE)

INTERVENTIONS:
Behavioral: Pregnant Body Project (PBP) — The Body Project is typically delivered as four 1-hour weekly sessions consisting of written, verbal, and behavioral exercises. The sessions aim to induce cognitive dissonance by encouraging participants to challenge the thin-ideal, a theoretically and empirically supported component of ED prevention. This adapted version of the Body Project (the Pregnant Body Project; PBP) consists of 6 1-hour, weekly group sessions delivered via Zoom. Since the target population consists of individuals with histories of an ED or disordered eating behaviors, PBP also includes elements from a treatment intervention (i.e., the Body Project Treatment 8.0 manual). PBP was adapted iteratively with a needs assessment, expert stakeholder input, and participant feedback following a mock trial with individuals with lived experience (i.e., individuals with histories of an ED who have given birth). This condition will be peer-delivered by facilitators with lived experience.
  Arms: Pregnant Body Project (PBP)
Behavioral: Pregnancy Health Education (PHE) — This time- dose- and attention- matched control condition accounts for the potential effects of time spent and support from group members and facilitators. Participants assigned to the PHE group will also be asked to attend 6, 1-hour, weekly group sessions via Zoom. During the sessions participants receive psychoeducation on body image and disordered eating during pregnancy but will not engage in any dissonance-inducing exercises. Participants will also receive lifestyle education specific to pregnancy (e.g., proper nutrition, sleep, physical activity), tied back to body image and disordered eating.
  Arms: Pregnancy Health Education (PHE)

SUMMARY:
The investigators aim to conduct a feasibility randomized controlled trial (RCT) of an eating disorder prevention program (The Body Project, adapted for pregnancy) versus a health education control among pregnant individuals with histories of an ED. The investigators will test the feasibility, implementation outcomes, and its preliminary effectiveness in reducing the risk of elevated disordered eating and body dissatisfaction during pregnancy and postpartum.

DETAILED DESCRIPTION:
The investigators aim to conduct a feasibility randomized controlled trial (RCT) of an eating disorder prevention program (The Body Project, adapted for pregnancy) versus a health education control among pregnant individuals with histories of an ED. The investigators will test the feasibility, implementation outcomes, and its preliminary effectiveness in reducing the risk of elevated disordered eating and body dissatisfaction during pregnancy and postpartum.

The investigators will aim to recruit N=60 pregnant individuals (in their first or second trimester) with histories of an ED. Both the intervention and active control consist of 6, weekly, 1-hour group sessions (6-8 participants per group) delivered over Zoom. There are four assessment points: pre-intervention, post-intervention, 3 months postpartum, and 6 months postpartum. Participants will complete online surveys at each assessment point and a post-intervention exit interview (active intervention only).

ELIGIBILITY:
Inclusion Criteria:

1. Within the first or second trimester of pregnancy at enrollment
2. 18 years or older
3. Able to provide informed consent
4. Endorse a self-reported history of an eating disorder or disordered eating behaviors
5. Are willing and able to comply with all group and study procedures
6. English fluency and literacy

Exclusion Criteria:

1. A diagnosis of bipolar or psychotic disorder, active mania or psychosis or substance abuse, an active eating disorder (active eating disorder symptomology informed by the Screening, Brief Intervention, and Referral to Treatment for Eating Disorders (SBIRT-ED) tool and clinician discretion), being at immediate risk of self-harm
2. Do not have access to a device with a camera

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Any birthing persons are eligible
Enrollment: 60 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | 0 weeks
  The investigators will consider the program feasible if the investigators meet recruitment targets (N=60).
Session attendance | 6 weeks
  The investigators will assess what percentage of enrolled participants complete 4 or more sessions. The benchmark will be > 50% of participants will complete 4 or more sessions.
Drop Out | 6 weeks
  The investigators will assess what percentage of enrolled participants complete post-test assessments. The benchmark will be > 50% of participants will complete the post-test surveys and interviews.
Client satisfaction questionnaire (CSQ-8) | 6 weeks
  Assesses participants' satisfaction with the intervention. Scores range from 8 to 32 with higher scores indicating greater satisfaction. The benchmark will be that at least 70% of participants will have scores over and above the midpoint in both the PBP and PHE groups.
Credibility and Expectancy Questionnaire (CEQ) | 0 weeks
  Assesses participants' perceptions that the treatment will work after learning about the study. The first three items measure credibility, and the latter three items measure expectancy. It is scored on a scale of 3-27 with higher scores indicating greater confidence in the treatment. The benchmark will be that at least 70% of participants will have scores over and above the midpoint in both the PBP and PHE groups.
Feasibility of data collection | Through the study completion, approximately 1 year depend on gestational at enrollment
  E.g.: The investigators will assess the feasibility of quantitative measures with the benchmark of no questionnaires fully missing in >25% of participants
Adapted Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), & Feasibility of Intervention Measure | 6 weeks
  Assesses acceptability, appropriateness, and feasibility of the intervention and Facilitators and Barriers to Participating. Acceptability, appropriateness, and feasibility subscales each consist of 4 items ranging from 1-5. Scores can be calculated by averaging the 4 items and range from 1-5. Higher scores indicate greater acceptability, appropriateness, and feasibility. The benchmark will be that at least 70% of participants will have scores over and above the midpoint for these subscales in both the PBP and PHE groups. Facilitators and Barriers to participating are open-ended questions and will be assessed with qualitative analyses.
Facilitator Adherence to Sessions | Through the study completion, approximately 1 year depend on gestational at enrollment
  The investigators will assess the percentage of sessions with ≥75% adherence. The benchmark will be ≥70% of sessions will have ≥75% adherence (checklist and audio recordings); 20% of sessions rated.
Participant Adherence to Homework | 6 weeks
  The investigators will assess the percentage of participants that complete (i.e., upload/submit) ≥75% of the homework assignments. The benchmark will be ≥70% of participants will complete ≥75% of the homework assignments.

SECONDARY OUTCOMES:
Thin Ideal Internalization Scale | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures the degree to which a person identifies with the notion that thinness is equivalent to attractiveness, with items ranging from 1-5. Scores are calculated by averaging the 8 items, and range from 1-5, with higher scores indicating greater internalization of the thin ideal.
Dutch Restrained Eating Scale | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures the frequency of dieting behaviors, with items ranging from 1-5. Scores are calculated by averaging the 10 items, and range from 1-5, with higher scores indicating increased levels of restrictive eating.
The Satisfaction and Dissatisfaction with Body Parts Scale | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures body dissatisfaction, with items ranging from 1-5. Scores are calculated by averaging the 9 items, and range from 1-5, with higher scores indicating greater body dissatisfaction.
Body Image in Pregnancy Scale (BIPS) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  36 items that measure body image during pregnancy, with items ranging from 1-5. The measure is made up of seven subscales: 'preoccupation with physical appearance' (six items), 'dissatisfaction with facial features' (four items), 'sexual attractiveness' (six items), 'prioritizing appearance over body functioning' (five items), 'appearance-related behavioral avoidance' (three items), and 'dissatisfaction with body parts' (six items). Subscale scores are calculated by averaging items, and range from 1-5, with higher scores indicating greater body image disturbance. The investigators adapted wording to administer the questionnaire again during postpartum.
Eating Disorder Examination Questionnaire (EDEQ) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  28-item questionnaire measuring ED psychopathology, with items ranging from 0-6. A global score is obtained by averaging all items except for 13-18, with higher scores indicating increased ED symptoms. The clinical cut-off score is 2.8, which indicates a probable ED. Items 13-18 assess frequency of ED behaviors and are not included in the global score.
Prenatal Eating Behaviors Screening (PEBS) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures ED psychopathology during pregnancy, with items ranging from 1-5. Scores are calculated by summing the 12 items, and range from 12-60, with higher scores indicating greater ED symptomatology during pregnancy. Scores >39 indicate a current ED.
Intuitive Eating Scale-3 (IES-3) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures intuitive eating, with items ranging from 1-5. A global score can be calculated by averaging the 12 items, and range from 1-5, with higher scores indicating greater levels of intuitive eating. Subscales (Unconditional Permission to Eat, Eating for Physical Reasons, Reliance on Hunger and Satiety Cues, and Body-Food Choice Congruence) can be calculated by averaging items specific to each subscale.
Eating Disorder Diagnostic Scale (EDDS) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Provides tentative diagnoses of full threshold anorexia nervosa, full threshold bulimia nervosa, full threshold binge eating disorder, subthreshold anorexia nervosa, subthreshold bulimia nervosa, and subthreshold binge eating disorder. The EDDS also generates an overall ED symptom score based on the sum of all relevant items. Higher scores indicate increased disorder eating symptomology with a clinical cut-off score of 16.5 for the overall symptom composite score (Krabbenborg et al., 2011).
  Krabbenborg, M. A., Danner, U. N., Larsen, J. K., van der Veer, N., van Elburg, A. A., de Ridder, D. T., Evers, C., Stice, E., & Engels, R. C. (2012). The Eating Disorder Diagnostic Scale: psychometric features within a clinical population and a cut-off point to differentiate clinical patients from healthy controls. European eating disorders review : the journal of the Eating Disorders Association, 20(4), 315-320. https://doi.org/10.1002/erv.1144
Edinburgh Postnatal Depression Scale (EPDS) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures depression in pregnancy and postpartum, with items ranging from 0-3. Scores are calculated by summing the 10 items, and range from 0-30, with higher scores indicating greater depressive symptoms.
Generalized Anxiety Disorder Assessment (GAD-7) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures anxiety, with items ranging from 0-3. Scores are calculated by summing the 7 items, and range from 0-21, with higher scores indicating greater anxiety.
Multidimensional Scale of Perceived Social Support (MSPSS) | 0 weeks, 6 weeks, 3 months pp, 6 months pp
  Measures perceived social support, with items ranging from 1-7. A global score is calculated by summing the 12 items, and ranges from 12-84, with higher scores indicating greater perceived social support. Subscales (Significant Other, Family, and Friends) can be calculated by averaging items specific to each subscale.
Participant Feedback | 6 weeks
  The investigators will conduct exit interviews with participants assigned to the PBP group. The investigators will use this to make further adaptations to the intervention. This is a qualitative assessment informed by the Consolidated Framework Implementation Research.
Facilitator Feedback | Through the intervention program completion, approximately 1 year
  The investigators will conduct exit interviews with the PBP group facilitators. The investigators will use this to make further adaptations to the intervention. This is not a scale. It is a survey including open test qualitative questions.
Neonatal Outcomes | 3 months pp
  Patient reported measures of infant health at birth (e.g., preterm birth, low birthweight), maternal and delivery complications (e.g., preeclampsia), provider interactions, pregnancy and postpartum experiences, and feeding experiences with their baby. Exploratory analyses and descriptive statistics will be conducted for these neonatal outcomes and pregnancy, postpartum and feeding experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Vanderkruik, PhD, MSc, Principal Investigator — The Center for Women's Mental Health at Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Vanderkruik R, Frisch CM, Woodworth EC, Scharner S, Bartels SJ, Freeman MP, Cohen LS, Stice E. The pregnant body project pilot RCT protocol: Preventing disordered eating behaviors in high-risk pregnant individuals. Contemp Clin Trials. 2025 Sep;156:108039. doi: 10.1016/j.cct.2025.108039. Epub 2025 Jul 31. PMID 40752822